CLINICAL TRIAL: NCT05726851
Title: A First-in-Human, Single Ascending Dose and Pharmacokinetic/Pharmacodynamic Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of Intravenous Infusions of E2025 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of E2025 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E2025-A001-001
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: E2025; Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A, Cohort 1: E2025 Dose 1 or Placebo (Experimental): Participants will receive E2025 Dose 1 or E2025 matching placebo (normal saline) administered as an IV infusion on Day 1.
  Interventions: Drug: E2025; Drug: Placebo
- Part A, Cohort 2: E2025 Dose 2 or Placebo (Experimental): Participants will receive E2025 Dose 2 or E2025 matching placebo (normal saline) administered as an IV infusion on Day 1.
  Interventions: Drug: E2025; Drug: Placebo
- Part A, Cohort 3: E2025 Dose 3 or Placebo (Experimental): Participants will receive E2025 Dose 3 or E2025 matching placebo (normal saline) administered as an IV infusion on Day 1.
  Interventions: Drug: E2025; Drug: Placebo
- Part A, Cohort 4: E2025 Dose 4 or Placebo (Experimental): Participants will receive E2025 Dose 4 or E2025 matching placebo (normal saline) administered as an IV infusion on Day 1.
  Interventions: Drug: E2025; Drug: Placebo
- Part B, Cohort 5: E2025 Dose 2 (Experimental): Participants will receive E2025 Dose 2 administered as an IV infusion on Day 1.
  Interventions: Drug: E2025
- Part B, Cohort 6: E2025 Dose 3 (Experimental): Participants will receive E2025 Dose 3 administered as an IV infusion on Day 1.
  Interventions: Drug: E2025
- Part B Cohort 7: E2025 Dose 4 (Experimental): Participants will receive E2025 Dose 4 administered as an IV infusion on Day 1.
  Interventions: Drug: E2025

INTERVENTIONS:
Drug: E2025 — E2025 IV infusion.
Drug: Placebo — E2025 matched placebo IV infusion.
  Arms: Part A, Cohort 1: E2025 Dose 1 or Placebo; Part A, Cohort 2: E2025 Dose 2 or Placebo; Part A, Cohort 3: E2025 Dose 3 or Placebo; Part A, Cohort 4: E2025 Dose 4 or Placebo

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of single intravenous (IV) infusions of E2025 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, male or female age greater than or equal to (>=) 18 years and less than or equal to (<=) 55 years old at the time of informed consent. Females must be of nonchildbearing potential
* Body weight >=50 kilogram (kg) and a Body Mass Index (BMI) >=18 and less than (<) 30 kilogram per square meter (kg/m^2) at Screening

Exclusion Criteria:

* Females who are breastfeeding or pregnant at Screening or Baseline; Females of childbearing potential.
* Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period or for 203 days after their partner's study drug administration.
* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
* Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
* Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening
* A prolonged QT/QTc interval (QTcF >450 millisecond [ms]). A history of risk factors for torsade de pointes or the use of concomitant medications that prolonged the QT/QTc interval
* Persistent systolic blood pressure (BP) greater than 130 millimeter of mercury (mmHg) or diastolic BP greater than 85 mmHg at Screening or Baseline; Heart rate less than 50 or more than 100 beats per minute at Screening or Baseline
* Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the Columbia-suicide Severity Rating Scale (C-SSRS) or equivalent scale or via interview with a psychiatrist
* Any lifetime history of psychiatric disease (including but not limited to depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, anxiety disorders); any current psychiatric symptoms as indicated by a standard screening tool.
* Known history of clinically significant drug allergy; known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
* Any history of hypersensitivity reaction to a foreign protein, with clinical features not limited to nasal or conjunctival symptoms such as in allergic rhinitis
* Known to be human immunodeficiency virus positive and/or active viral hepatitis (hepatitis B core antibody [HBcAb], hepatitis B viral protein [HBcAg], hepatitis B surface antigen [HBsAg], hepatitis C virus antibody [HCVAb]) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within the 2 years before Screening, or a positive urine drug test or breath alcohol test at Screening or Baseline
* Currently enrolled in another clinical study or used any investigational drug or device within 28 days (or 5*the half-life, whichever is longer) preceding informed consent
* Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
* Exposure to any biologic drug within 90 days or at least 5 half-lives (whichever is longer), or within 4 weeks for vaccines, before Screening, with the exception of flu (7 days before dosing) and COVID-19 vaccination (14 days before dosing until after the Follow-up visit).
* Any contraindication to continuous CSF sampling via indwelling lumbar catheter or via lumbar puncture (LP)
* Participants identified at risk for hemorrhage.
* Inadequate venous access that would interfere with study drug administration or obtaining blood samples
* Participants who contravene the restrictions on concomitant medications, food, beverages, physical activities, and others as defined in the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Screening up to Day 113
Number of Participants With Clinically Significant Abnormal Laboratory Values | Screening up to Day 113
Number of Participants With Clinically Significant Abnormal Vital Signs Values | Screening up to Day 113
Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs) Findings | Screening up to Day 113
Number of Participants With Clinically Significant Abnormal Physical Examinations Findings | Screening up to Day 113
Number of Participants With Clinically Significant Abnormal Psychiatric Examination Findings | Screening up to Day 8

SECONDARY OUTCOMES:
Cmax: Maximum Observed Serum Concentration for E2025 | Day 1: 0-24 hours up to Day 113
Tmax: Time to Reach Maximum Observed Serum Concentration (Cmax) for E2025 | Day 1: 0-24 hours up to Day 113
AUC(0-t): Area Under the Serum Concentration-time Curve From Time Zero to Last Quantifiable Concentration for E2025 | Day 1: 0-24 hours up to Day 113
AUC(0-inf): Area Under the Serum Concentration-time Curve From Time Zero to Infinite for E2025 | Day 1: 0-24 hours up to Day 113
AUC(0-24h): Area Under the Serum Concentration-time Curve From Time Zero to 24 hours for E2025 | Day 1: 0-24 hours
AUC(0-72h): Area Under the Serum Concentration-time Curve From Time Zero to 72 hours for E2025 | Day 1: 0-72 hours
AUC(0-672h): Area Under the Serum Concentration-time Curve From Time Zero to 672 hours for E2025 | Day 1: 0-672 hours
t1/2: Terminal Elimination Phase Half-life for E2025 | Day 1: 0-24 hours up to Day 113
CL/F: Apparent Total Clearance for E2025 | Day 1: 0-24 hours up to Day 113
Vss: Volume of Distribution at Steady State for E2025 | Day 1: 0-24 hours up to Day 113
Part A: Cerebrospinal Fluid (CSF) Concentrations for E2025 | Pre-dose; Days 8 and 29 post-dose
Part B, CSF Cmax: Maximum Observed CSF Concentration for E2025 | Day 1: 0-24 hours up to Day 99
Part B, CSF Tmax: Time to Reach Maximum Observed CSF Concentration (Cmax) for E2025 | Day 1: 0-24 hours up to Day 99
Part B, CSF AUC(0-24h): Area Under the CSF Concentration-time Curve From Time Zero to 24 hours for E2025 | Day 1: 0-24 hours
Part B: Ratio of Cmax in CSF and Cmax in Serum for E2025 | Day 1: 0-24 hours up to Day 99
Part B: Ratio of AUC(0-24h) in CSF and AUC(0-24h) in Serum for E2025 | Day 1: 0-24 hours
Serum Concentration of Anti- E2025 Antibodies | Day 1 up to Day 113

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.